CLINICAL TRIAL: NCT05097573
Title: Clinical Evaluation of the Efficacy of Fractional Radiofrequency for the Treatment and Reduction of Stretch Marks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI0119
Record Dates: First submitted 2021-10-04; First posted 2021-10-28 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Stretch Mark
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Venus Viva (Experimental): The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids, stretch marks and scars. Beginning with the Baseline visit (Visit 1), subjects will receive a total of 4 treatments approximately 4 weeks apart.
  Interventions: Device: Venus Viva

INTERVENTIONS:
Device: Venus Viva — The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, stretch marks, rhytids and scars. Beginning with the Baseline visit (Visit 1), subjects will receive a total of 4 treatments approximately 4 weeks apart.

SUMMARY:
This is a prospective, single centre, evaluator-blind study of the performance of fractional radiofrequency (RF) for the treatment and revision of stretch marks. The study will evaluate the progress of 15 subjects requesting treatment of stretch marks. The study will involve four treatments on both sides of the face with 4 week intervals between each treatment. Subjects will be followed at 12 and 16 weeks after their last treatment. Analysis will be performed on all subjects who receive at least one treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects, 18-60 years of age who are seeking treatment for their stretch marks
2. Fitzpatrick skin type I-IV
3. Able to read, understand and voluntarily provide written Informed Consent.
4. Able and willing to comply with the treatment/follow-up schedule and requirements.

Exclusion Criteria:

1. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body (e.g. cochlear implant).
2. Subjects with any implantable metal device in the treatment area
3. Permanent implant in the treated area, such as metal plates and screws (excluding dental implants), or an injected chemical substance.
4. Current or history of any kind of cancer, or dysplastic nevi in the treated area.
5. Severe concurrent conditions, such as cardiac disorders.
6. Impaired immune system due to immunosuppressive diseases, such as AIDS and HIV, or use of immunosuppressive medications.
7. History of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area; may be enrolled only following a prophylactic regime.
8. Poorly controlled endocrine disorders, such as diabetes.
9. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
10. History of skin disorders, such as keloids, abnormal wound healing, as well as very dry and fragile skin.
11. History of bleeding coagulopathies, or use of anticoagulants.
12. Use of isotretinoin (Accutane®) or other systemic retinoids limited up to 10mg/day or as per investigators discretion.
13. Treating over tattoo or permanent makeup.
14. Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Skinpulse Dermatologie, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Venus Viva
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Venus Viva
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick skin type (or phototype) describes a way to classify the skin by its reaction to exposure to sunlight. It is based on the amount of melanin in in the skin. Darker skin is a higher category. The PI evaluated the subjects' skin and categorized into a Fitzpatrick skin type. A person's Fitzpatrick score is set and does not change.
  Participants
    I | 1
    II | 10
    III | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Volume of Striae Via Antera 3D Imaging System Analysis From Baseline to 16 Weeks Post-final Treatment
Description: Change from baseline to the follow-up visit 16 weeks post-final treatment as a percentage of baseline volume.
Time Frame: 16 Weeks Post-Final Treatment (Week 28)
Measure: Mean (Standard Error); unit: percentage change from baseline
Units Other Than Participants: striae sites on the body
Arm/Group | Venus Viva
Number analyzed (Participants) | 15
Number analyzed (striae sites on the body) | 55
percentage change from baseline | -28.3 (4.7)

2. Primary Outcome: Overall Stretch Mark Improvement From Baseline to 16 Weeks Post-Final Treatment Assessed by the Global Aesthetic Improvement Scale (GAIS)
Description: Evaluate the efficacy of overall stretch mark improvement assessed live by the Investigator and a subject assessment of stretch mark including the Global Aesthetic Improvement Scale (GAIS).The Global Aesthetic Improvement Scale is a seven-grade subjective test. The PI evaluated before and after photographs and graded them for change.
  Possible responses were (3) Very Much Improved, (2) Much Improved, (1) Improved, (0) No Change, (-1) Worse, (-2) Much Worse, and (-3) Very Much Worse. For reporting of outcomes, the higher the GAIS value, the greater the improvement (Range -3 to 3).
Time Frame: 16 Weeks Post-Final Treatment (Week 28)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Venus Viva
Number analyzed (Participants) | 15
units on a scale | 1.7 (0.4)

3. Secondary Outcome: Subject Satisfaction
Description: Subjects' assessment of satisfaction with the treatment using a 5 point Subject Satisfaction Scale at 16 weeks post-treatment. The Subject Satisfaction Scale is a five-grade subjective test.
  Participants were asked to rate their satisfaction level with the results. Possible responses were (4) Very Satisfied, (3) Satisfied, (2) Having No Opinion, (1) Unsatisfied, and (0) Very Unsatisfied.
Time Frame: 16 Weeks Post-Final Treatment (Week 28)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Venus Viva
Number analyzed (Participants) | 15
units on a scale | 3.1 (0.3)

4. Secondary Outcome: Subject Scale - Visual Analog Scale for Pain
Description: Subject's assessment of discomfort and pain after treatments as measured by a 10 cm visual analog scale (VAS). The Visual Analog Scale is a scale from 0 cm (no pain) and 10 cm (pain as bad as it can be). Possible responses were of 0 to 0.4 cm can be considered (no pain); 0.5 to 4.4 cm (mild pain), 4.5 to 7.4 cm (moderate pain), and 7.5 to 10 cm (severe pain). No anaesthetic was used.
  An average of all 4 treatments was taken for each subject.
Time Frame: Treatment 1 (Week 1), Treatment 2 (Week 4), Treatment 3 (Week 8), Treatment 4 (Week 12)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Venus Viva
Number analyzed (Participants) | 17
units on a scale | 3.8 (0.2)

5. Secondary Outcome: Subject Scale - 5 Point Scale for Treatment Tolerability
Description: Subject's assessment of treatment tolerability as measured by a 5-point scale. Participants were asked about their tolerability level immediately post-treatment. Possible scores were; (4) Very Tolerable, (3) Tolerable, (2) Having No Opinion, (1) Intolerable, and (0) Very Intolerable.
  An average of all 4 treatments was taken for each subject.
Time Frame: Treatment 1 (Week 1), Treatment 2 (Week 4), Treatment 3 (Week 8), Treatment 4 (Week 12)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Venus Viva
Number analyzed (Participants) | 17
units on a scale | 3.1 (0.2)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Venus Viva
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venus Viva (N=17)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT05097573/Prot_000.pdf